CLINICAL TRIAL: NCT07226570
Title: Central Neural Actions of Ibogaine in Opioid Use Disorder (OUD)
Brief Title: Mapping Ibogaine Neural Dynamics in Opioid Use Disorder
Acronym: MIND-OUD
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Richard Edmund Harris, Professor, University of California, Irvine
Other Study IDs: 7038
Record Dates: First submitted 2025-10-22; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder (OUD)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults (21-65) with Opioid Use Disorder Receiving Ibogaine
  Interventions: Other: Observational study with MRI/EEG

INTERVENTIONS:
Other: Observational study with MRI/EEG — Participants will independently undergo ibogaine treatment at a licensed clinic outside the United States. The UCI research team will not provide the ibogaine treatment but will conduct observational imaging and qualitative assessments before and after. These include MRI and MRS scans to measure brain activity and chemistry, EEG recordings of brain wave activity, urine toxicology and pregnancy tests, and self-report questionnaires on craving, withdrawal, mood, pain, anxiety, and quality of life.

SUMMARY:
This study aims to understand how ibogaine treatment may change brain activity and symptoms in people with moderate-severe opioid use disorder (OUD), as defined by the DSM-5. Ibogaine is a plant-derived compound that some studies suggest can reduce opioid cravings and withdrawal. Participants in this study will already be independently scheduled to receive legal ibogaine treatment at a licensed clinic outside of the U.S. The University of California, Irvine (UCI) research team will not provide the treatment but will conduct brain imaging, administer psychometric questionnaires, and obtain urine samples throughout the course of this study.

The main goal is to see if ibogaine changes brain function as assessed with magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS), and electroencephalography (EEG). MRI/MRS will measure brain activity when participants view opioid-related images, brain connectivity at rest, and levels of brain chemicals involved in craving and substance use. EEG will measure brain wave activity. MRI/MRS/EEG will be administered across 3 study time points. In addition, participants will complete psychometric surveys related to opioid craving, withdrawal symptoms, mood, anxiety, pain, and quality of life, along with urine tests to monitor substance use and screen for pregnancy.

The investigators hypothesize that after ibogaine treatment, participants will show reduced brain responses to opioid cues, changes in brain connectivity and chemistry, and improvements in self-reported cravings and other symptoms. This information may help researchers better understand how ibogaine works in the brain and whether it could play a role in future treatments for OUD.

DETAILED DESCRIPTION:
Primary Hypothesis:

3-5 days and 1-month after ibogaine treatment (compared to baseline), participants will show reduced brain responses to opioid-related images on task fMRI and reduced resting-state connectivity within reward circuitry. The brain areas expected to be affected include the basal ganglia, cingulate cortex, hippocampus, and amygdala. Post-ibogaine spectroscopy will also show lower glutamate + glutamine (Glx) levels within the insula and nucleus accumbens.

Exploratory Hypotheses:

The magnitude of MRI/MRS changes (including activation/connectivity in the cingulate, hippocampus, and amygdala) will correlate with improvements in opioid craving and related symptoms measured by validated questionnaires (e.g., VAS craving, SOWS, CEQ).

EEG will show relative increases in alpha power, relative decreases in gamma power, and decreases in frontal alpha frequency and signal complexity, which will track with reductions in craving and withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21-65 with confirmed moderate to severe OUD as assessed by equal or greater than 4 symptoms using DSM-5 criteria.
* Independently scheduled to receive ibogaine treatment at a licensed clinic outside the U.S.
* Able to undergo MRI and EEG procedures at UC Irvine at Visit 1 (baseline), Visit 4, and Visit 5, totaling three sessions.
* Able to complete psychometric surveys at each study time point.
* Able to provide urine samples at all three scanning sessions, as well as 3- and 6-month follow-ups.
* Able to independently coordinate transportation to UC Irvine at 3- and 6-month follow-up visits.
* Capable of giving written informed consent.
* Proficient ability to speak, read, and write in English.

Exclusion Criteria:

* Presence of known past procedures, devices in the body, claustrophobia, or other contraindications for MRI.
* Use of any psychedelic substances within 3 months prior to screening.
* Diagnosis of schizophrenia, bipolar disorder (type I or II), or borderline personality disorder.
* Prior use of ibogaine.
* Pregnant or nursing. Participants who become pregnant during the study will be withdrawn from further participation.
* Diagnosis of epilepsy or history of seizures.
* Other contraindications to MRI/EEG methods. These may include but are not limited to: brain surgical clips and surgical staples, metal implants in the brain, and certain metallic dental material.
* Inability to complete MRI/EEG sessions or follow-up visits.
* Inability or unwillingness of an individual to give written informed consent.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ages 21 to 65 with a confirmed diagnosis of moderate to severe opioid use disorder (OUD), defined as meeting four or more symptoms according to DSM-5 criteria. Participants must be independently scheduled to receive ibogaine treatment at a licensed clinic outside the United States.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Resting-State Functional Connectivity in Reward Circuitry | Baseline (Visit 1; within 2 weeks of consent) and follow-up assessments approximately 4 to 6 weeks after baseline (Visits 4 and 5).
  Resting-state functional MRI will assess functional connectivity within reward circuitry, including the basal ganglia, nucleus accumbens, cingulate cortex, hippocampus, insula, and amygdala. Connectivity will be quantified using correlation coefficients between regional BOLD signals.
  Unit of Measure: Correlation coefficient (range: -1 to +1, where higher values indicate stronger positive connectivity)
Change in BOLD Activation to Drug Cues During Task-Based fMRI | Baseline (Visit 1; within 2 weeks of consent) and follow-up assessments approximately 4 to 6 weeks after baseline (Visits 4 and 5).
  Task-based functional MRI will measure blood-oxygen-level-dependent (BOLD) signal activation in reward-related brain regions (basal ganglia, nucleus accumbens, cingulate cortex, hippocampus, insula, and amygdala) while participants view opioid-related versus neutral images.
  Unit of Measure: Percent signal change in BOLD activation
Change in Glutamate+Glutamine Concentration in Nucleus Accumbens | Baseline (Visit 1; within 2 weeks of consent) and follow-up assessments approximately 4 to 6 weeks after baseline (Visits 4 and 5).
  Proton Magnetic Resonance Spectroscopy (1H-MRS) will measure glutamate+glutamine (Glx) concentration in the nucleus accumbens.
  Unit of Measure: Institutional units (ratio relative to creatine)
Change in Glutamate+Glutamine Concentration in Anterior Insula | Baseline (Visit 1; within 2 weeks of consent) and follow-up assessments approximately 4 to 6 weeks after baseline (Visits 4 and 5).
  Proton Magnetic Resonance Spectroscopy (1H-MRS) will measure glutamate+glutamine (Glx) concentration in the anterior insula.
  Unit of Measure: Institutional units (ratio relative to creatine)

SECONDARY OUTCOMES:
Change in Resting-State EEG Alpha Band Power | Baseline (Visit 1; within 2 weeks of consent) and follow-up assessments approximately 4 to 6 weeks after baseline (Visits 4 and 5).
  Electroencephalography (EEG) will be recorded using a 64-electrode BrainVision system during resting-state conditions. Alpha band power (8-12 Hz) will be quantified from averaged spectral analysis.
  Unit of Measure: Microvolts squared (μV²)
Change in Subjective Opiate Withdrawal Scale (SOWS) Score | Baseline to end of study (8.5 months)
  The Subjective Opiate Withdrawal Scale (SOWS) is a self-report questionnaire, typically with 16 items, designed to measure the severity of common opiate withdrawal symptoms experienced by individuals. Each item asks the respondent to rate the severity of a specific withdrawal symptom on a scale, allowing for a quantified subjective experience of withdrawal.
  Unit of Measure: Score on a scale (0-64, higher = greater withdrawal intensity)
Change in Opioid Craving Visual Analog Scale (OC-VAS) Score | Baseline to end of study (8.5 months)
  The Opioid Craving Visual Analog Scale is a self-report measure used to assess the subjective intensity of opioid craving. Participants indicate their current level of craving by marking a point along a 100 mm line anchored at each end with "no craving" (0) and "extreme craving" (100). The distance from the "no craving" anchor to the participant's mark represents the craving score. Higher scores indicate greater craving intensity (i.e., worse outcome).
  Unit of Measure: Score on a scale (0-100, higher = worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Harris, PhD, Principal Investigator — University of California, Irvine, Susan Samueli Integrative Health Institute
Locations (1):
- Susan Samueli Integrative Health Institute, University of California, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Drug Overdose Data — https://www.cdc.gov/nchs/nvss/vsrr/drug-overdose-data.htm